CLINICAL TRIAL: NCT02749552
Title: The Role of Values, Acceptance, and Mindfulness Strategies in Long Term Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3168
Record Dates: First submitted 2016-04-08; First posted 2016-04-25 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acceptance and Commitment Therapy (Experimental): ACT intervention
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — weight-related interventions using values, acceptance, and mindfulness based on Acceptance and Commitment Therapy

SUMMARY:
Obesity is a prevalent, destructive, and costly chronic disease. In 2008, 37% of Canadian adults were measured as overweight, and 25% as obese. Obesity is a risk factor for a number of serious health problems, including type 2 diabetes, asthma, gallbladder disease, osteoarthritis, chronic back pain, several types of cancers (i.e., colorectal, kidney, breast, endometrial, ovarian and pancreatic cancers) and cardiovascular disease (i.e., hypertension, stroke, congestive heart failure and coronary artery disease). In 2008, it was estimated that the annual economic burden of obesity in Canada was $4.6 billion. Given the economic strain and widespread health risks of obesity, there is a clear need to provide effective interventions for obesity.

The purpose of the proposed study is to examine the role of ACT-based interventions in long-term weight maintenance. The proposed study will examine the role of value consistent behaviour, acceptance skills, and mindfulness skills in promoting long-term weight-related health behaviours. Acceptance and Commitment Therapy (ACT) is an empirically supported psychological intervention that emphasizes value consistent behaviours, acceptance skills and mindfulness skills.

DETAILED DESCRIPTION:
Participants will be recruited from the weight loss surgery waitlist and randomly assigned to a brief (5 sessions) ACT intervention or to waitlist control group. A mobile app will be used to encourage daily ACT skill practice and track health behaviours over time. The primary objective of the proposed project is to test whether a brief ACT intervention can result in sustained weight management (at 6 months and 1 year) compared to a waitlist control group. If this brief format of ACT intervention for obesity proves to be effective in encouraging health behaviours and weight loss, it may provide a low cost, sustainable option to enhance much needed obesity management services in Nova Scotia.

ELIGIBILITY:
Inclusion Criteria:

* BMI above 30 who are participating in Weight Loss Surgery program at the Nova Scotia Health Authority

Exclusion Criteria:

* None

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
health behaviours (self-report questionnaires) | 5 years
  engagement in weight related health behaviours (i.e., dietary choices)
health behaviours (self-report questionnaires) | 5 years
  engagement in weight related health behaviours (i.e., physical activity)

SECONDARY OUTCOMES:
acceptance (self-report questionnaire) | 5 years
  ability to acknowledge and tolerate distressing thoughts, feelings, and sensations (total score is used)
mindfulness (self-report questionnaire) | 5 years
  ability to engage in purposeful, present-moment awareness

CONTACTS AND LOCATIONS:
Overall Officials: Dayna Lee-Baggley, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Weight Loss Surgery - Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lillis J, Hayes SC, Bunting K, Masuda A. Teaching acceptance and mindfulness to improve the lives of the obese: a preliminary test of a theoretical model. Ann Behav Med. 2009 Feb;37(1):58-69. doi: 10.1007/s12160-009-9083-x. Epub 2009 Feb 28. PMID 19252962
- [Background] Forman EM, Butryn ML. A new look at the science of weight control: how acceptance and commitment strategies can address the challenge of self-regulation. Appetite. 2015 Jan;84:171-80. doi: 10.1016/j.appet.2014.10.004. Epub 2014 Oct 16. PMID 25445199